CLINICAL TRIAL: NCT00181948
Title: A Pilot Study of Strattera Treatment in Children With Attention-Deficit/Hyperactivity Disorder Who Have Poor Response to Stimulant Therapy
Brief Title: Strattera Treatment in Children With ADHD Who Have Poor Response to Stimulant Therapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Joseph Biederman, MD, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2004-P-000883
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2010-06-22 (Estimated); Status verified 2010-06

CONDITIONS: ADHD
Keywords: ADHD; children; stimulant non-responders; Strattera
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Atomoxetine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: atomoxetine (Strattera)

SUMMARY:
This will be a 6-week, unblinded study using the medication Strattera for children and adolescents with attention deficit hyperactivity disorder (ADHD) who failed to respond to an adequate trial of stimulant treatment. Specific hypotheses are as follows:

Hypothesis 1: ADHD symptomatology in youth with ADHD will be responsive to Strattera treatment in the short term.

Hypothesis 2: Strattera treatment (in doses of up to 120 mg/day or 1.2 mg/kg/day) in children and adolescents with ADHD will be safe and well tolerated.

DETAILED DESCRIPTION:
Strattera (atomoxetine) is a non-stimulant presynaptic norepinephrine reuptake inhibitor recently approved by the Food and Drug Administration for use in child, adolescent and adult patients with ADHD. Atomoxetine is a potent inhibitor of the presynaptic norepinephrine transporter with minimal affinity for other noradrenergic receptors or for other neurotransmitter transporters or receptors. Thus, Strattera could be a viable alternative treatment for ADHD individuals who do not respond to stimulants.

The purpose of this study is to assess the effectiveness, safety and tolerability of Strattera in youth, ages 6-17 years with ADHD who failed to respond to an adequate trial of stimulant treatment. If this initial study shows proof of the concept, we will follow-up the study with a randomized clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Male and female outpatients 6-17 years of age.
* Subjects with the diagnosis of attention deficit hyperactivity disorder (ADHD), by the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV), as manifested in clinical evaluation and confirmed by structured interview.
* ADHD rating scale-symptom checklist > 24
* Subjects with a past history of depression, bipolar disorder, anxiety disorder (including obsessive compulsive disorder [OCD]) without current disorder for > 3 months as ascertained through structured diagnostic interview and clinical exam.
* Subjects treated for anxiety disorders and depression (with non-MAOI antidepressants [e.g., SSRIs, bupropion, venlafaxine] or benzodiazepines) who are on a stable medication regimen for at least three months, and who have a disorder specific Clinical Global Impression (CGI)-severity score ≤ 3 (mildly ill) and who have a score on the Hamilton-Depression and Hamilton-Anxiety Rating Scale below 15 (mild range) will be included in the study.
* Subjects with a past or present history of tics will be eligible.
* Subjects with a past history of substance use disorders but drug and alcohol free for > 6 months.
* Subjects with mild cases of asthma and allergy will be included.
* Potential subjects will have failed an adequate trial of a stimulant as defined by:

  * Subjects who had intolerable side effects on a stimulant, or
  * Poor response (an ADHD CGI-I of > 3) on at least 4 weeks of > 1.0 mg/kg/day of a methylphenidate product; or > 0.5 mg/kg/day of an amphetamine product.
* Only English-speaking subjects will be allowed into the study for the following reasons:

  1. the assessment instruments are not available and have not been adequately standardized in other languages;
  2. the clinical trials facility is located in Cambridge and not in the Massachusetts General Hospital (MGH) main campus without the availability of translators;
  3. psychiatric questionnaires and evaluations are taxing and adding the complexity of a translator has the potential to make the patient experience even more exhausting.

Exclusion Criteria:

* Any clinically unstable psychiatric conditions including the following:

  * acute psychosis,
  * acute panic,
  * acute OCD,
  * acute mania,
  * acute suicidality,
  * acute substance use disorders (alcohol or drugs),
  * sociopathy,
  * criminality.
* Any metabolic, neurological, hepatic, renal, cardiovascular, hematological, ophthalmic, or endocrine disease.
* Clinically significant abnormal baseline laboratory values which include the following:

  * Values which deviate greater than 20% from the normal ranges of the laboratory standard for a basic metabolic screen and complete blood count.
  * Exclusionary blood pressure parameters will include any values above 140 (systolic) and 90 (diastolic).
  * Exclusionary electrocardiogram (ECG) parameters will include a QTC > 460 msec, QRS >120 msec, and PR > 200 msec. Subjects having ECG evidence of ischemia or arrhythmia as reviewed by an independent cardiologist.
* Mental retardation (intelligence quotient [I.Q.] < 75).
* Organic brain disorders.
* Seizures.
* Pregnant or nursing females.
* Subjects with current adequate treatment for ADHD or a history of a previous adequate trial of Strattera.
* Prior hypersensitivity to atomoxetine.
* MAOI antidepressant use currently or within two weeks of starting study.
* Urinary retention or bladder dysfunction.
* Narrow angle glaucoma.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2004-09; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Symptom reduction using Clinical Global Impression (ADHD) | administered weekly
ADHD Symptom Checklist | administered weekly

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Biederman, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Cambridge, Massachusetts, United States